CLINICAL TRIAL: NCT03888066
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized Withdrawal, Parallel Group Study of Patiromer for the Management of Hyperkalemia in Subjects Receiving Renin Angiotensin Aldosterone System Inhibitor (RAASi) Medications for the Treatment of Heart Failure (DIAMOND)
Brief Title: Patiromer for the Management of Hyperkalemia in Subjects Receiving RAASi Medications for the Treatment of Heart Failure (DIAMOND)
Acronym: DIAMOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PAT-CR-302; 2018-005030-38 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-25 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Hyperkalemia
Keywords: treatment of hyperkalemia; chronic kidney disease; hypertension; hyperkalemia; potassium; spironolactone; heart failure; Renin Angiotensin-Aldosterone System Inhibitor (RAASi); RAASi; high potassium; eplerenone; reduced ejection fraction
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic; Hypertension; Heart Failure | interventions — patiromer

STUDY DESIGN:
Intervention Model Description: Prospective Phase 3b multinational, multicenter, double-blind, placebo-controlled, randomized withdrawal, parallel group study that includes screening and 12 weeks Run-in Phase and a randomized withdrawal Blinded Treatment Phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Patiromer (Experimental): Subjects will be randomized to receive a daily dose of patiromer with possible dose adjustments based on subsequent local serum potassium levels.
  Interventions: Drug: Patiromer
- Group 2: Placebo (Placebo Comparator): Subjects will be randomized to receive a daily dose of placebo with possible dose adjustments based on subsequent local serum potassium levels.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Patiromer — The starting dose of patiromer will be 1 packet/day and may be taken either with food or without food. Based upon the patiromer treatment algorithm patiromer may be increased by 1 packet per day in intervals of at least 1 week (± 3 days). For subjects who become hypokalemic, patiromer may be decreased to a minimum of 0 packets/day. Doses of patiromer will be 0 packets/day, 1 packet/day, 2 packets/day, and 3 packets/day (maximum dose).
  Other Names: Veltassa
  Arms: Group 1: Patiromer
Drug: Placebos — The starting dose of placebo will be 1 packet/day and may be taken either with food or without food. Based upon the placebo treatment algorithm placebo may be increased by 1 packet per day in intervals of at least 1 week (± 3 days). For subjects who become hypokalemic, placebo may be decreased to a minimum of 0 packets/day. Doses of placebo will be 0 packets/day, 1 packet/day, 2 packets/day, and 3 packets/day (maximum dose).
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to assess the effects of patiromer compared with placebo on serum K+ in HF patients.

DETAILED DESCRIPTION:
Prospective Phase 3b multinational, multicenter, double-blind, placebo-controlled, randomized withdrawal, parallel group study that includes screening and up to 12 weeks Run-in Phase (all subjects will have patiromer initiated and RAASi medications, including mineralocorticoid receptor antagonist (MRA) optimized) and a randomized withdrawal Blinded Treatment Phase.

The study population includes subjects with heart failure (HF) with reduced ejection fraction (HFrEF) who are hyperkalemic (serum potassium [K+] > 5.0 mEq/L) while receiving treatment with renin angiotensin aldosterone system inhibitor (RAASi) medications or who are normokalemic (serum K+ 4.0 - 5.0 mEq/L) but have a history of hyperkalemia prior to screening with subsequent reduction or discontinuation of a RAASi medication.

Each subject's participation includes a Run-in Phase (maximum 12 weeks) followed by the Treatment Phase (variable per subject). Study duration for individual subjects will vary, depending on their individual enrollment date. Subjects who prematurely discontinue patiromer/placebo will remain in the study for the collection of clinical events data and will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years or greater
* Symptomatic low ejection fraction heart failure (weak heart muscle)
* Receiving any dose of a beta blocker for the treatment of HF (unless not able to tolerate)
* Kidney function not more than mild or moderately impaired
* High blood potassium (>5.0 mEq/L) currently while receiving medications for heart failure OR normal blood potassium currently but previously had high potassium in the12 months prior to screening which caused a permanent reduction or discontinuation of heart failure medications
* Hospitalization for heart failure or treatment in an out patient setting with intravenous medications within the last 12 months before screening.

Exclusion Criteria:

* Current acute decompensated HF, within 4 weeks before screening. Subjects with a discharge from a hospitalization for acute decompensation of HF longer than 4 weeks before screening may be included
* Significant primary aortic or mitral valvular heart disease (except secondary mitral regurgitation due to left ventricular dilatation)
* Heart transplantation or planned heart transplantation (i.e., currently on a heart transplant waiting list) during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1195 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szecsödy, MD, Study Director — Vifor Pharma
Locations (415):
- United States (133):
  - Investigator Site 11-080, Alexander City, Alabama
  - Investigator Site 11-041, Huntsville, Alabama
  - Investigator Site 11-153, Phoenix, Arizona
  - Investigator Site 11-097, Tucson, Arizona
  - Investigator Site 11-052, Bakersfield, California
  - Investigator Site 11-174, Fremont, California
  - Investigator Site 11-136, Fresno, California
  - Investigator Site 11-102, Huntington Beach, California
  - Investigator Site 11-162, La Jolla, California
  - Investigator Site 11-048, La Mesa, California
  - Investigator Site 11-111, Laguna Hills, California
  - Investigator Site 11-017, Long Beach, California
  - Investigator Site 11-128, Northridge, California
  - Investigator Site 11-035, Pasadena, California
  - Investigator Site 11-044, Sacramento, California
  - Investigator Site 11-135, San Diego, California
  - Investigator Site 11-086, San Diego, California
  - Investigator Site 11-112, Santa Ana, California
  - Investigator Site 11-101, Stockton, California
  - Investigator Site 11-047, Thousand Oaks, California
  - Investigator Site 11-057, Van Nuys, California
  - Investigator Site 11-058, West Hills, California
  - Investigator Site 11-095, Aurora, Colorado
  - Investigator Site 11-168, Altamonte Springs, Florida
  - Investigator Site 11-106, Boynton Beach, Florida
  - Investigator Site 11-028, Brandon, Florida
  - Investigator Site 11-003, Doral, Florida
  - Investigator Site 11-138, Gainesville, Florida
  - Investigator Site 11-164, Greenacres City, Florida
  - Investigator Site 11-078, Homestead, Florida
  - Investigator Site 11-004, Jacksonville, Florida
  - Investigator Site 11-179, Jacksonville, Florida
  - Investigator Site 11-122, Medley, Florida
  - Investigator Site 11-115, Miami, Florida
  - Investigator Site 11-125, Miami, Florida
  - Investigator Site 11-005, Miami, Florida
  - Research Site 11-001, Miami Lakes, Florida
  - Research Site 11-002, Miami Lakes, Florida
  - Investigator Site 11-032, North Miami Beach, Florida
  - Investigator Site 11-171, Orlando, Florida
  - Investigator Site 11-025, Orlando, Florida
  - Investigator Site 11-087, Orlando, Florida
  - Investigator Site 11-177, Pembroke Pines, Florida
  - Investigator Site 11-144, Pompano Beach, Florida
  - Investigator Site 11-099, Tamarac, Florida
  - Investigator Site 11-090, Tampa, Florida
  - Investigator Site 11-163, Tampa, Florida
  - Investigator Site 11-109, Atlanta, Georgia
  - Investigator Site 11-015, Columbus, Georgia
  - Investigator Site 11-141, Macon, Georgia
  - Investigator Site 11-031, Arlington Heights, Illinois
  - Investigator Site 11-051, Hazel Crest, Illinois
  - Investigator Site 11-063, Peoria, Illinois
  - Investigator Site 11-137, Peoria, Illinois
  - Investigator Site 11-117, Merrillville, Indiana
  - Investigator Site 11-129, Munster, Indiana
  - Investigator Site 11-069, Richmond, Indiana
  - Investigator Site 11-061, Owensboro, Kentucky
  - Investigator Site 11-183, Opelousas, Louisiana
  - Investigator Site 11-022, West Monroe, Louisiana
  - Investigator Site 11-027, Baltimore, Maryland
  - Investigator Site 11-023, Columbia, Maryland
  - Investigator Site 11-132, Boston, Massachusetts
  - Investigator Site 11-123, Detroit, Michigan
  - Investigator Site 11-121, Livonia, Michigan
  - Investigator Site 11-076, Rochester, Michigan
  - Investigator Site 11-189, Rochester, Michigan
  - Investigator Site 11-068, Jackson, Mississippi
  - Investigator Site 11-154, Kansas City, Missouri
  - Investigator Site 11-094, St Louis, Missouri
  - Investigator Site 11-071, Lincoln, Nebraska
  - Investigator Site 11-049, Las Vegas, Nevada
  - Investigator Site 11-145, North Las Vegas, Nevada
  - Investigator Site 11-088, Haddon Heights, New Jersey
  - Investigator Site 11-054, Linden, New Jersey
  - Investigator Site 11-148, New Brunswick, New Jersey
  - Investigator Site 11-107, Newark, New Jersey
  - Investigator Site 11-116, Albuquerque, New Mexico
  - Investigator Site 11-151, Brooklyn, New York
  - Investigator Site 11-126, Brooklyn, New York
  - Investigator Site 11-073, Buffalo, New York
  - Investigator Site 11-040, Manhasset, New York
  - Investigator Site 11-053, Richmond Hill, New York
  - Investigator Site 11-081, Staten Island, New York
  - Investigator Site 11-021, Stony Brook, New York
  - Investigator Site 11-127, The Bronx, New York
  - Investigator Site 11-120, Charlotte, North Carolina
  - Investigator Site 11-075, Charlotte, North Carolina
  - Investigator Site 11-018, Greenville, North Carolina
  - Investigator Site 11-157, Lumberton, North Carolina
  - Investigator Site 11-149, Columbus, Ohio
  - Investigator Site 11-064, Lorain, Ohio
  - Investigator Site 11-042, Marion, Ohio
  - Investigator Site 11-187, Toledo, Ohio
  - Investigator Site 11-074, Bartlesville, Oklahoma
  - Investigator Site 11-124, Oklahoma City, Oklahoma
  - Investigator Site 11-056, Hillsboro, Oregon
  - Investigator Site 11-169, Portland, Oregon
  - Investigator Site 11-165, Erie, Pennsylvania
  - Investigator Site 11-082, Hershey, Pennsylvania
  - Investigator Site 11-110, Greenville, South Carolina
  - Investigator Site 11-098, Greenwood, South Carolina
  - Investigator Site 11-119, Lancaster, South Carolina
  - Investigator Site 11-133, Rock Hill, South Carolina
  - Investigator Site 11-152, Chattanooga, Tennessee
  - Investigator Site 11-091, Jackson, Tennessee
  - Investigator Site 11-142, Memphis, Tennessee
  - Investigator Site 11-083, Memphis, Tennessee
  - Investigator Site 11-134, Tullahoma, Tennessee
  - Investigator Site 11-104, Allen, Texas
  - Investigator Site 11-185, Allen, Texas
  - Investigator Site 11-070, Amarillo, Texas
  - Investigator Site 11-176, Dallas, Texas
  - Investigator Site 11-092, Dallas, Texas
  - Investigator Site 11-170, Denison, Texas
  - Investigator Site 11-060, Fort Worth, Texas
  - Investigator Site 11-072, Gonzales, Texas
  - Investigator Site 11-140, Houston, Texas
  - Investigator Site 11-089, Houston, Texas
  - Investigator Site 11-146, Houston, Texas
  - Investigator Site 11-156, Houston, Texas
  - Investigator Site 11-034, Katy, Texas
  - Investigator Site 11-029, Lampasas, Texas
  - Investigator Site 11-046, McKinney, Texas
  - Investigator Site 11-147, San Antonio, Texas
  - Investigator Site 11-085, San Antonio, Texas
  - Investigator Site 11-161, Sugar Land, Texas
  - Investigator Site 11-160, Webster, Texas
  - Investigator Site 11-178, Salt Lake City, Utah
  - Investigator Site 11-158, Norfolk, Virginia
  - Investigator Site 11-188, Norfolk, Virginia
  - Investigator Site 11-065, Morgantown, West Virginia
  - Investigator Site 11-045, Milwaukee, Wisconsin
- Argentina (17):
  - Investigator Site 21-006, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Investigator Site 21-007, Ciudadela, Buenos Aires
  - Investigator Site 21-019, Mar del Plata, Buenos Aires
  - Investigator Site 21-020, Ramos Mejía, Buenos Aires
  - Investigator Site 21-004, San Nicolás de los Arroyos, Buenos Aires
  - Investigator Site 21-011, Córdoba, Córdoba Province
  - Investigator Site 21-021, Córdoba, Córdoba Province
  - Investigator Site 21-014, Córdoba, Córdoba Province
  - Investigator Site 21-015, Villa María, Córdoba Province
  - Investigator Site 21-010, San Miguel de Tucumán, Tucumán Province
  - Investigator Site 21-012, Buenos Aires
  - Investigator Site 21-003, Buenos Aires
  - Investigator Site 21-018, Buenos Aires
  - Investigator Site 21-008, Buenos Aires
  - Investigator Site 21-017, Salta
  - Investigator Site 21-005, San Luis
  - Investigator Site 21-009, Santa Fe
- Belgium (10):
  - Investigator Site 44-002, Mechelen, Antwerp
  - Investigator Site 44-001, Ghent, Oost Vlaanderen
  - Investigator Site 44-005, Aalst
  - Investigator Site 44-009, Brussels
  - Investigator Site 44-003, Genk
  - Investigator Site 44-008, Hasselt
  - Investigator Site 44-007, Leuven
  - Investigator Site 44-006, Liège
  - Investigator Site 44-010, Roeselare
  - Investigator Site 44-004, Yvoir
- Brazil (23):
  - Investigator Site 22-019, Fortaleza, Ceará
  - Investigator Site 22-013, Fortaleza, Ceará
  - Investigator Site 22-012, Vitória, Espírito Santo
  - Investigator Site 22-021, Salvador, Estado de Bahia
  - Investigator Site 22-023, Brasília, Federal District
  - Investigator Site 22-011, Belo Horizonte, Minas Gerais
  - Investigator Site 22-005, Belo Horizonte, Minas Gerais
  - Investigator Site 22-004, Uberlândia, Minas Gerais
  - Investigator Site 22-010, Campina Grande do Sul, Paraná
  - Investigator Site 22-008, Canoas, Rio Grande do Sul
  - Investigator Site 22-003, Porto Alegre, Rio Grande do Sul
  - Investigator Site 22-015, Porto Alegre, Rio Grande do Sul
  - Investigator Site 22-002, Porto Alegre, Rio Grande do Sul
  - Investigator Site 22-009, Porto Alegre, Rio Grande do Sul
  - Investigator Site 22-025, Porto Alegre, Rio Grande do Sul
  - Investigator Site 22-017, Blumenau, Santa Catarina
  - Investigator Site 22-007, Aracaju, Sergipe
  - Investigator Site 22-016, Campinas, São Paulo
  - Investigator Site 22-018, Ribeirão Preto, São Paulo
  - Investigator Site 22-020, São José do Rio Preto, São Paulo
  - Investigator Site 22-024, Rio de Janeiro
  - Investigator Site 22-014, São Paulo
  - Investigator Site 22-022, São Paulo
- Bulgaria (8):
  - Investigator Site 61-003, Burgas
  - Investigator Site 61-002, Pleven
  - Investigator Site 61-004, Plovdiv
  - Investigator Site 61-010, Rousse
  - Investigator Site 61-009, Sofia
  - Investigator Site 61-008, Sofia
  - Investigator Site 61-005, Sofia
  - Investigator Site 61-006, Sofia
- Canada (9):
  - Investigator Site 12-005, Winnipeg, Manitoba
  - Investigator Site 12-013, St. John's, Newfoundland and Labrador
  - Investigator Site 12-008, Cambridge, Ontario
  - Investigator Site 12-012, London, Ontario
  - Investigator Site 12-010, Newmarket, Ontario
  - Investigator Site 12-002, Toronto, Ontario
  - Investigator Site 12-009, Greenfield Park, Quebec
  - Investigator Site 12-006, Sherbrooke, Quebec
  - Investigator Site 12-004, Trois-Rivières, Quebec
- Czechia (13):
  - Investigator Site 62-004, Bílina
  - Investigator Site 62-019, Brno
  - Investigator Site 62-017, Havířov
  - Investigator Site 62-005, Havlíčkův Brod
  - Investigator Site 62-013, Liberec
  - Investigator Site 62-015, Litovel
  - Investigator Site 62-010, Mariánské Lázně
  - Investigator Site 62-018, Náchod
  - Investigator Site 62-001, Prague
  - Investigator Site 62-012, Prague
  - Investigator Site 62-009, Prague
  - Investigator Site 62-011, Slaný
  - Investigator Site 62-016, Uherské Hradiště
- France (20):
  - Investigator Site 32-010, Bordeaux
  - Investigator Site 32-002, La Tronche
  - Investigator Site 32-014, Lille
  - Investigator Site 32-020, Lyon
  - Investigator Site 32-005, Montpellier
  - Investigator Site 32-001, Nancy
  - Investigator Site 32-004, Paris
  - Investigator Site 32-008, Paris
  - Investigator Site 32-017, Paris
  - Investigator Site 32-007, Paris
  - Investigator Site 32-003, Pau
  - Investigator Site 32-015, Poitiers
  - Investigator Site 32-013, Reims
  - Investigator Site 32-019, Rouen
  - Investigator Site 32-018, Saint-Brieuc
  - Investigator Site 32-006, Toulon
  - Investigator Site 32-012, Toulouse
  - Investigator Site 32-009, Tourcoing
  - Investigator Site 32-011, Valenciennes
  - Investigator Site 32-016, Valenciennes
- Georgia (12):
  - Investigator Site 63-012, Batumi
  - Investigator Site 63-007, Tbilisi
  - Investigator Site 63-011, Tbilisi
  - Investigator Site 63-004, Tbilisi
  - Investigator Site 63-002, Tbilisi
  - Investigator Site 63-006, Tbilisi
  - Investigator Site 63-008, Tbilisi
  - Investigator Site 63-010, Tbilisi
  - Investigator Site 63-003, Tbilisi
  - Investigator Site 63-009, Tbilisi
  - Investigator Site 63-001, Tbilisi
  - Investigator Site 63-005, Tbilisi
- Germany (23):
  - Investigator Site 33-011, Coburg, Bavarian
  - Investigator Site 33-008, Greifswald, Mecklenburg-Vorpommern
  - Investigator Site 33-006, Homburg, Saarland
  - Investigator Site 33-023, Bad Oeynhausen
  - Investigator Site 33-020, Berlin
  - Investigator Site 33-013, Berlin
  - Investigator Site 33-015, Bielefeld
  - Investigator Site 33-016, Bremen
  - Investigator Site 33-004, Erfurt
  - Investigator Site 33-001, Essen
  - Investigator Site 33-019, Frankfurt
  - Investigator Site 33-007, Frankfurt
  - Investigator Site 33-018, Giessen
  - Investigator Site 33-002, Halle
  - Investigator Site 33-005, Hamburg
  - Investigator Site 33-022, Hanover
  - Investigator Site 33-012, Heilbronn
  - Investigator Site 33-017, Kiel
  - Investigator Site 33-021, Leipzig
  - Investigator Site 33-010, Leverkusen
  - Investigator Site 33-024, Minden
  - Investigator Site 33-014, Nuremberg
  - Investigator Site 33-003, Würzburg
- Hungary (7):
  - Investigator Site 64-010, Budapest
  - Investigator Site 64-002, Budapest
  - Investigator Site 64-006, Budapest
  - Investigator Site 64-009, Budapest
  - Investigator Site 64-001, Kecskemét
  - Investigator Site 64-007, Kistarcsa
  - Investigator Site 64-005, Nyíregyháza
- Israel (14):
  - Investigator Site 35-008, Ashkelon
  - Investigator Site 35-009, Be’er Ya‘aqov
  - Investigator Site 35-003, Hadera
  - Investigator Site 35-006, Haifa
  - Investigator Site 35-007, Haifa
  - Investigator Site 35-002, Holon
  - Investigator Site 35-005, Jerusalem
  - Investigator Site 35-014, Jerusalem
  - Investigator Site 35-001, Jerusalem
  - Investigator Site 35-010, Nahariya
  - Investigator Site 35-011, Petah Tikva
  - Investigator Site 35-013, Ramat Gan
  - Investigator Site 35-012, Safed
  - Investigator Site 35-016, Tiberias
- Italy (11):
  - Investigator Site 34-005, Ancona
  - Investigator Site 34-002, Bergamo
  - Investigator Site 34-007, Brescia
  - Investigator Site 34-001, Caserta
  - Investigator Site 34-009, Cona
  - Investigator Site 34-014, Foggia
  - Investigator Site 34-010, Genova
  - Investigator Site 34-004, Milan
  - Investigator Site 34-012, Piacenza
  - Investigator Site 34-003, Roma
  - Investigator Site 34-013, San Bonifacio
- Mexico (9):
  - Investigator Site 23-012, Guadalajara, Jalisco
  - Investigator Site 23-004, Guadalajara, Jalisco
  - Investigator Site 23-007, Cuauhtémoc, Mexico City
  - Investigator Site 23-005, Gustavo Adolfo Madero, Mexico City
  - Investigator Site 23-010, San Pedro Garza García, Nuevo Léon
  - Investigator Site 23-011, Oaxaca City, Oaxaca
  - Investigator Site 23-001, Querétaro City, Querétaro
  - Investigator Site 23-002, Culiacán, Sinaloa
  - Investigator Site 23-006, Xalapa, Veracruz
- Netherlands (13):
  - Investigator Site 36-003, Rotterdam, South Holland
  - Investigator Site 36-002, 's-Hertogenbosch
  - Investigator Site 36-012, Amstelveen
  - Investigator Site 36-006, Blaricum
  - Investigator Site 36-009, Dirksland
  - Investigator Site 36-015, Dordrecht
  - Investigator Site 36-007, Ede
  - Investigator Site 36-001, Groningen
  - Investigator Site 36-013, Helmond
  - Investigator Site 36-014, Hoorn
  - Investigator Site 36-010, Schiedam
  - Investigator Site 36-004, Tilburg
  - Investigator Site 36-011, Utrecht
- Poland (14):
  - Investigator Site 65-007, Bialystok
  - Investigator Site 65-014, Katowice
  - Investigator Site 65-012, Kędzierzyn-Koźle
  - Investigator Site 65-001, Lodz
  - Investigator Site 65-018, Lodz
  - Investigator Site 65-019, Olsztyn
  - Investigator Site 65-015, Ostrowiec Świętokrzyski
  - Investigator Site 65-021, Pomorskie
  - Investigator Site 65-003, Poznan
  - Investigator Site 65-020, Poznan
  - Investigator Site 65-008, Rzeszów
  - Investigator Site 65-010, Wroclaw
  - Investigator Site 65-005, Wroclaw
  - Investigator Site 65-011, Zgierz
- Russia (17):
  - Investigator Site 66-014, Izhevsk, Udmurt Republic
  - Investigator Site 66-008, Chelyabinsk
  - Investigator Site 66-016, Kazan'
  - Investigator Site 66-010, Kemerovo
  - Investigator Site 66-015, Moscow
  - Investigator Site 66-004, Moscow
  - Investigator Site 66-011, Moscow
  - Investigator Site 66-017, Moscow
  - Investigator Site 66-002, Novosibirsk
  - Investigator Site 66-005, Penza
  - Investigator Site 66-007, Perm
  - Investigator Site 66-012, Petrozavodsk
  - Investigator Site 66-018, Ryazan
  - Investigator Site 66-013, Saint Petersburg
  - Investigator Site 66-003, Saint Petersburg
  - Investigator Site 66-009, Tver'
  - Investigator Site 66-001, Yekaterinburg
- Serbia (8):
  - Investigator Site 67-010, Belgrade
  - Investigator Site 67-002, Belgrade
  - Investigator Site 67-004, Belgrade
  - Investigator Site 67-008, Belgrade
  - Investigator Site 67-001, Kamenitz
  - Investigator Site 67-005, Niš
  - Investigator Site 67-007, Niška Banja
  - Investigator Site 67-003, Šabac
- Spain (25):
  - Investigator Site 37-014, Palma de Mallorca, Balearic Islands
  - Investigator Site 37-010, Castellon, Castellon
  - Investigator Site 37-003, Barcelona, Catalonia
  - Investigator Site 37-005, Santiago de Compostela, La Coruña
  - Investigator Site 37-011, Majadahonda, Madrid
  - Investigator Site 37-024, Marbella, Malaga
  - Investigator Site 37-016, San Cristóbal de La Laguna, Tenerife
  - Investigator Site 37-001, Manises, Valencia
  - Investigator Site 37-025, A Coruña
  - Investigator Site 37-012, Alicante
  - Investigator Site 37-015, Badalona
  - Investigator Site 37-007, Barcelona
  - Investigator Site 37-002, Barcelona
  - Investigator Site 37-018, Huelva
  - Investigator Site 37-023, Lleida
  - Investigator Site 37-004, Madrid
  - Investigator Site 37-006, Madrid
  - Investigator Site 37-021, Madrid
  - Investigator Site 37-020, Madrid
  - Investigator Site 37-026, Madrid
  - Investigator Site 37-017, Málaga
  - Investigator Site 37-022, Murcia
  - Investigator Site 37-013, Seville
  - Investigator Site 37-009, Valencia
  - Investigator Site 37-008, Valencia
- Ukraine (17):
  - Investigator Site 68-008, Kharkiv, Novobavarskiy
  - Investigator Site 68-017, Dnipro
  - Investigator Site 68-009, Ivano-Frankivsk
  - Investigator Site 68-005, Ivano-Frankivsk
  - Investigator Site 68-001, Kharkiv
  - Investigator Site 68-011, Kharkiv
  - Investigator Site 68-010, Kharkiv
  - Investigator Site 68-002, Kharkiv
  - Investigator Site 68-012, Kyiv
  - Investigator Site 68-003, Kyiv
  - Investigator Site 68-015, Kyiv
  - Investigator Site 68-013, Kyiv
  - Investigator Site 68-007, Kyiv
  - Investigator Site 68-006, Lviv
  - Investigator Site 68-014, Vinnytsia
  - Investigator Site 68-016, Zaporizhzhya
  - Investigator Site 68-004, Zhytomyr
- United Kingdom (12):
  - Investigator Site 39-012, Harlow, Essex
  - Investigator Site 39-003, Scunthorpe, North Lincolshire
  - Investigator Site 39-005, Dudley, West Midlands
  - Investigator Site 39-009, Barnsley
  - Investigator Site 39-016, High Wycombe
  - Investigator Site 39-008, Inverness
  - Investigator Site 39-011, Leicester
  - Investigator Site 39-013, Liverpool
  - Investigator Site 39-015, London
  - Investigator Site 39-010, North Shields
  - Investigator Site 39-007, Swansea
  - Investigator Site 39-004, York

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later.
  Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and the study sponsor and researchers must sign a data sharing agreement.

REFERENCES:
- [Derived] Coats AJS, Anker SD, Lund LH, Filippatos G, Rossignol P, Pitt B, Weir MR, Kosiborod MN, Metra M, Bohm M, Ezekowitz JA, Bayes-Genis A, Mentz RJ, Ponikowski P, Senni M, Cleland JGF, Goudev A, Khintibidze I, Lindenfeld J, Merkely B, Waechter S, Budden J, Perrin A, Butler J. Patiromer for Heart Failure Medication Optimization in Patients With Current or Past Hyperkalemia: DIAMOND Subanalysis. JACC Heart Fail. 2024 Dec;12(12):2026-2037. doi: 10.1016/j.jchf.2024.08.003. Epub 2024 Sep 25. PMID 39340493
- [Derived] Butler J, Anker SD, Lund LH, Coats AJS, Filippatos G, Siddiqi TJ, Friede T, Fabien V, Kosiborod M, Metra M, Pina IL, Pinto F, Rossignol P, van der Meer P, Bahit C, Belohlavek J, Bohm M, Brugts JJ, Cleland JGF, Ezekowitz J, Bayes-Genis A, Gotsman I, Goudev A, Khintibidze I, Lindenfeld J, Mentz RJ, Merkely B, Montes EC, Mullens W, Nicolau JC, Parkhomenko A, Ponikowski P, Seferovic PM, Senni M, Shlyakhto E, Cohen-Solal A, Szecsody P, Jensen K, Dorigotti F, Weir MR, Pitt B. Patiromer for the management of hyperkalemia in heart failure with reduced ejection fraction: the DIAMOND trial. Eur Heart J. 2022 Nov 1;43(41):4362-4373. doi: 10.1093/eurheartj/ehac401. PMID 35900838
- [Derived] Bolanos JA, Seliger SL. Recurrent Hyperkalemia in Renin-Angiotensin-Aldosterone System Inhibitor (RAASi) Treatment: Stuck between a Rock and a Hard Place. Clin J Am Soc Nephrol. 2021 Mar 8;16(3):345-347. doi: 10.2215/CJN.00950121. Epub 2021 Feb 19. No abstract available. PMID 33608263

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From a total of 1642 screened participants, 1195 entered the Run-in Phase. The Run-in Phase Set includes participants who signed the informed consent and received at least 1 dose of patiromer during the Run-in Phase but were not eligible to be randomized. A total of 1168 participants received patiromer during Run-in Phase, and 878 of these participants were randomized to receive patiromer or placebo during the Treatment Phase
Groups:
- Patiromer: Randomized participants who received a daily dose of patiromer, with possible dose adjustments based on subsequent local serum potassium level, during the Treatment Phase.
  The starting dose of patiromer was 1 packet/day taken either with food or without food. Based upon the K+ management algorithms, patiromer was to be increased by 1 packet per day in intervals of at least 1 week (±3 days). If hypokalemia developed during the Treatment Phase, then the study drug was to be down titrated (lowest acceptable dose was 0 packets/day) until local serum K+ ≥4.0 mEq/l. Doses of patiromer were 0 packets/day, 1 packet/day, 2 packets/day, and 3 packets/day (maximum dose).
  mEq/l = Milliequivalents Per Liter
- Placebo: Randomized participants who received a daily dose of placebo, with possible dose adjustments based on subsequent local serum potassium level, during the Treatment Phase.
  The starting dose of placebo was 1 packet/day taken either with food or without food. Based upon the K+ management algorithms, placebo was to be increased by 1 packet per day in intervals of at least 1 week (±3 days). If hypokalemia developed during the Treatment Phase, then the study drug was to be down-titrated (lowest acceptable dose was 0 packets/day) until local serum K+ ≥4.0 mEq/l. Doses of placebo were 0 packets/day, 1 packet/day, 2 packets/day, and 3 packets/day (maximum dose).
  mEq/l = Milliequivalents Per Liter
Period: Run-in Phase
Arm/Group | Patiromer | Placebo
Started | 1195 | 0
Completed | 878 | 0
Not Completed | 317 | 0
Not completed — Randomization Criterion #1 | 24 | 0
Not completed — Randomization Criteria #1, #2 | 5 | 0
Not completed — Randomization Criteria #1, #2 #4; AE; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — Randomization Criteria #1, #3 | 1 | 0
Not completed — Randomization Criteria #1, #4 | 1 | 0
Not completed — Randomization Crit #1, #4; Withdraw By Subject; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — Randomization Criteria #1, #4; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — Randomization Criterion #1; AE | 4 | 0
Not completed — Randomization Criterion #1; AE; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — Randomization Criterion #1; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 2 | 0
Not completed — Randomization Criterion #2 | 5 | 0
Not completed — Randomization Criteria #2, #3 | 1 | 0
Not completed — Randomization Criteria #2, #3, #4 | 1 | 0
Not completed — Randomization Criteria #2, #4 | 4 | 0
Not completed — Randomization Criterion #3 | 11 | 0
Not completed — Randomization Criteria #3, #4 | 1 | 0
Not completed — Randomization Criteria #3, #4; 2 Wks After Taking Min 0 Packet/Day, sK+ Is < 4.0 Meq/L | 2 | 0
Not completed — Randomization Criterion #3; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — Randomization Criterion #4 | 3 | 0
Not completed — Randomization Criterion #3; Physician Decision | 1 | 0
Not completed — Randomization Criterion #4; AE | 4 | 0
Not completed — Randomization Criterion #4; AE; 2 Wks After Taking Min 0 Packet/Day, sK+ Is < 4.0 Meq/L | 1 | 0
Not completed — Randomization Criterion #3; Exceeded 12 Weeks Of Run In | 1 | 0
Not completed — Randomization Criterion #4; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 2 | 0
Not completed — Randomization Criterion #4; 2 Wks After Taking Min 0 Packet/Day, sK+ Is < 4.0 Meq/L | 1 | 0
Not completed — AE (Adverse Event) | 17 | 0
Not completed — AE; Withdrawal By Subject | 3 | 0
Not completed — AE; Withdrawal By Subject; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — AE; 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 1 | 0
Not completed — AE; 2 Wks After Taking Min 0 Packet/Day, sK+ Is < 4.0 Meq/L | 2 | 0
Not completed — Withdrawal by Subject | 43 | 0
Not completed — AE; Physician Decision | 1 | 0
Not completed — 1 Wk After 3 Patiromer Packets/Day, sK+ >5.0 Meq/L | 10 | 0
Not completed — Withdrawal By Subject; Withdrawal Of Consent | 1 | 0
Not completed — 2 Wks After Taking Min 0 Packet/Day, sK+ Is < 4.0 Meq/L | 6 | 0
Not completed — Death | 1 | 0
Not completed — Non-Compliance With Study Drug | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 13 | 0
Not completed — Sponsor Request | 34 | 0
Not completed — Study Terminated By Sponsor | 71 | 0
Not completed — Withdrawal Of Consent | 1 | 0
Not completed — Exceeded 12 Weeks Of Run In | 2 | 0
Not completed — Not treated with Patiromer during Run-in | 27 | 0
Period: Treatment Phase (Overall Study)
Arm/Group | Patiromer | Placebo
Started | 439 | 439
Completed | 360 | 367
Not Completed | 79 | 72
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 20 | 13
Not completed — Adverse Event | 27 | 21
Not completed — Lost to Follow-up | 1 | 0
Not completed — Consent withdrawn by subject | 21 | 25
Not completed — End of study visit not completed/delayed | 1 | 3
Not completed — Early study termination | 0 | 1
Not completed — Treatment discontinuation | 2 | 2
Not completed — Delayed visit and insufficient study | 6 | 6
Not completed — Sponsor's decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patiromer: Randomized participants who received a daily dose of patiromer, with possible dose adjustments based on subsequent local serum potassium level, during the Treatment Phase.
  The starting dose of patiromer was 1 packet/day taken either with food or without food. Based upon the K+ management algorithms, patiromer was to be increased by 1 packet per day in intervals of at least 1 week (±3 days). If hypokalemia developed during the Treatment Phase, then the study drug was to be down titrated (lowest acceptable dose was 0 packets/day) until local serum K+ ≥4.0 mEq/l. Doses of patiromer were 0 packets/day, 1 packet/day, 2 packets/day, and 3 packets/day (maximum dose).
- Placebo: Randomized participants who received a daily dose of placebo, with possible dose adjustments based on subsequent local serum potassium level, during the Treatment Phase.
  The starting dose of placebo was 1 packet/day taken either with food or without food. Based upon the K+ management algorithms, placebo was to be increased by 1 packet per day in intervals of at least 1 week (±3 days). If hypokalemia developed during the Treatment Phase, then the study drug was to be down-titrated (lowest acceptable dose was 0 packets/day) until local serum K+ ≥4.0 mEq/l. Doses of placebo were 0 packets/day, 1 packet/day, 2 packets/day, and 3 packets/day (maximum dose).
- Total: Total of all reporting groups
Arm/Group | Patiromer | Placebo | Total
Number analyzed (Participants) | 439 | 439 | 878
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 181 | 169 | 350
  >=65 years | 258 | 270 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.0) | 67.1 (9.9) | 66.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 126 | 238
  Male | 327 | 313 | 640
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 57 | 113
  Not Hispanic or Latino | 381 | 379 | 760
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Argentina | 16 | 16 | 32
  Belgium | 0 | 2 | 2
  Brazil | 6 | 10 | 16
  Bulgaria | 43 | 48 | 91
  Canada | 1 | 0 | 1
  Czechia | 2 | 7 | 9
  France | 1 | 1 | 2
  Georgia | 139 | 118 | 257
  Germany | 4 | 2 | 6
  Hungary | 8 | 11 | 19
  Israel | 8 | 4 | 12
  Italy | 3 | 4 | 7
  Mexico | 6 | 4 | 10
  Netherlands | 3 | 1 | 4
  Poland | 37 | 43 | 80
  Russia | 37 | 42 | 79
  Serbia | 3 | 5 | 8
  Spain | 11 | 14 | 25
  Ukraine | 81 | 75 | 156
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum K+ Levels From Baseline
Description: Adjusted mean changes in serum K+ from Baseline.
Time Frame: Mean duration of exposure: 227.9 days for Patiromer and 234.5 days for Placebo
Measure: Least Squares Mean (Standard Error); unit: Milliequivalents Per Liter (mEq/l)
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 439 | 439
Milliequivalents Per Liter (mEq/l) | 0.029 (0.019) | 0.127 (0.019)
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Difference in adjusted mean changes (SE); Test type: Superiority; p < 0.001, Mixed model for repeated measures (MMRM); Mean Difference (Final Values) = -0.097, 95% CI 2-sided [-0.128 to -0.067], Standard Error of Mean 0.015

2. Secondary Outcome: CIF Estimates of the Time to First Hyperkalemia Event With Serum K+ Level > 5.5 mEq/l Over Time
Description: Cumulative incidence of the first event of hyperkalemia with a serum K+ value >5.5 mEq/l taking death as competing and calculated as CIF Estimates (95% CI) over time.
  Aalen-Johansen estimators of the cumulative incidence function with death as a competing event.
  CIF = cumulative incidence function; mEq/l = Milliequivalents Per Liter
Time Frame: From Day 1/Baseline to week 90
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 439 | 439
Probability
  Week 1 | 0.02 [0.01 to 0.04] | 0.04 [0.03 to 0.06]
  Week 2 | 0.04 [0.02 to 0.06] | 0.08 [0.06 to 0.11]
  Week 6 | 0.05 [0.03 to 0.07] | 0.10 [0.08 to 0.13]
  Week 18 | 0.08 [0.06 to 0.12] | 0.14 [0.11 to 0.18]
  Week 30 | 0.13 [0.10 to 0.17] | 0.20 [0.15 to 0.24]
  Week 42 | 0.17 [0.12 to 0.22] | 0.24 [0.19 to 0.29]
  Week 54 | 0.21 [0.15 to 0.27] | 0.29 [0.23 to 0.35]
  Week 66 | 0.25 [0.18 to 0.32] | 0.34 [0.26 to 0.42]
  Week 78 | 0.30 [0.22 to 0.40] | 0.34 [0.26 to 0.42]
  Week 90 | 0.34 [0.23 to 0.44] | 0.34 [0.26 to 0.42]
Statistical Analysis 1: Comparison: Patiromer vs Placebo; Hazard Ratio patiromer vs placebo. The HR for the time to first hyperkalemia event for patiromer vs placebo was calculated. HR and p-value come from a Cox proportional regression model adjusted for geographic region, sex, Baseline T2DM status, Baseline K+ value, and Baseline eGFR. HR = Hazard Ratio; T2DM=Type 2 diabetes mellitus; eGFR=Estimated glomerular filtration rate; Test type: Superiority; p = 0.006, Regression, Cox — Threshold for statistical significance = 0.05; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.45 to 0.87]

3. Secondary Outcome: CIF Estimates of the Reduction of the MRA Dose Below Target Dose Over Time
Description: Cumulative incidence of the reduction of the MRA dose below target dose calculated as CIF Estimates (95% CI) over time.
  Note: The reduction below the MRA target dose must last for at least 14 days (orless if at the end of study) to confirm this endpoint.
  CIF = cumulative incidence function; mEq/l = Milliequivalents Per Liter
Time Frame: From Day 1/Baseline to week 102
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 439 | 439
Probability
  Week 1 | 0.02 [0.01 to 0.04] | 0.04 [0.03 to 0.07]
  Week 2 | 0.03 [0.02 to 0.05] | 0.08 [0.06 to 0.11]
  Week 6 | 0.06 [0.04 to 0.08] | 0.12 [0.09 to 0.15]
  Week 18 | 0.10 [0.08 to 0.14] | 0.15 [0.12 to 0.19]
  Week 30 | 0.14 [0.10 to 0.18] | 0.19 [0.15 to 0.23]
  Week 42 | 0.16 [0.12 to 0.21] | 0.23 [0.18 to 0.28]
  Week 54 | 0.19 [0.14 to 0.24] | 0.26 [0.20 to 0.32]
  Week 66 | 0.22 [0.16 to 0.29] | 0.27 [0.21 to 0.33]
  Week 78 | 0.27 [0.20 to 0.35] | 0.29 [0.22 to 0.36]
  Week 90 | 0.27 [0.20 to 0.35] | 0.29 [0.22 to 0.36]
  Week 102 | 0.27 [0.20 to 0.35] | NA [0 to 0] — Not feasible to estimate the cumulative incidence at a time beyond the largest observed time
Statistical Analysis 1: Comparison: Patiromer vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.006, Regression, Cox — Threshold for statistical significance = 0.05; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.45 to 0.87]

4. Secondary Outcome: Investigator-reported Events of Hyperkalemia
Description: Participant's follow-up is from the date of the first dose of randomized study medication up to the participant's end of study date or 24 Jun 2021, whichever comes first.
  Annualized event rate per 100 subject-years= The total number of events for all subjects in the treatment group divided by the total subject-years of follow-up in that treatment group multiplied by 100.
Time Frame: Mean duration of exposure: 227.9 days for Patiromer and 234.5 days for Placebo
Measure: Number; unit: Ann. event rate per 100 subject-years
Arm/Group | Patiromer | Placebo
Number analyzed (Participants) | 439 | 439
Ann. event rate per 100 subject-years | 82.38 | 114.65
Statistical Analysis 1: Comparison: Patiromer vs Placebo; NBMAC Annualized event RR patiromer vs placebo. NBMAC adjusted for geographical region, sex, Baseline T2DM status, Baseline K+ value, and Baseline eGFR. Rate ratio less than 1 favors patiromer. NBMAC=Negative binomial model adjusted for covariates; RR=Rate Ratio; T2DM=Type 2 diabetes mellitus; eGFR=Estimated glomerular filtration rate; Test type: Superiority; p < 0.001, Negative binomial model adjusted for cov; Annualized event rate ratio = 0.658, 95% CI 2-sided [0.534 to 0.81]

5. Secondary Outcome: Hyperkalemia-related Hard Outcomes Endpoints
Description: Analyzed using Win Ratio approach with the following hierarchical components:
  1. Time to CV death
  2. Total number of CV hospitalizations
  3. Total number of hyperkalemia toxicity events with serum K+ >6.5 mEq/l
  4. Total number of hyperkalemia events with serum K+ >6.0-6.5 mEq/l
  5. Total number of hyperkalemia events with serum K+ >5.0 mEq/l
  MHTE=More hyperkalemia toxicity events; MHE=More hyperkalemia events; CV=Cardiovascular
Time Frame: Mean duration of exposure: 227.9 days for Patiromer and 234.5 days for Placebo
Measure: Number; unit: Events
Groups:
- All Participants: All participants randomized to patiromer or placebo arm.
Arm/Group | All Participants
Number analyzed (Participants) | 878
Events
  CV death in Placebo Group First | 3491
  CV death in Patiromer Group First | 4609
  More CV hospitalizations in Placebo Group | 4539
  More CV hospitalizations in Patiromer Group | 4178
  MHTE with serum K+>6.5 in Placebo Group | 419
  MHTE with serum K+>6.5 in Patiromer Group | 401
  MHE with serum K+>6.0-6.5 in Placebo Group | 4283
  MHE with serum K+>6.0-6.5 in Patiromer Group | 1446
  MHE with serum K+>5.0-6.0 in Placebo Group | 55633
  MHE with serum K+>5.0-6.0 in Patiromer Group | 34156
  None of the above | 79566
  Total number of pairs | 192721
Statistical Analysis 1: Comparison: All Participants; Win ratio for composite. Win ratio approach: Patients in the new treatment and control groups are formed into matched pairs based on their risk profiles. For each matched pair, the new treatment patient is labelled winner/loser depending on CV/hyperkalemia event first. The win ratio is the total number of winners divided by the total numbers of losers; Test type: Superiority; p < 0.001, Win Ratio; Win Ratio = 1.526, 95% CI 2-sided [1.231 to 1.906]
Statistical Analysis 2: Comparison: All Participants; Win ratio CV death and hospitalization. Win ratio approach: Patients in the new treatment and control groups are formed into matched pairs based on their risk profiles. For each matched pair, the new treatment patient is labelled winner/loser depending on CV/hyperkalemia event first. The win ratio is the total number of winners divided by the total numbers of losers. Unmatched win ratio is presented for this endpoint. Win ratio above 1 favors patiromer; Test type: Superiority; p = 0.744, Win Ratio; Win Ratio = 0.914, 95% CI 2-sided [0.526 to 1.578]

6. Secondary Outcome: RAASi Use Score
Description: RAASi use score (0 to 8 points) analyzed using the Win Ratio approach for each pair of participants with the following additive components:
  1. All-cause death
  2. Occurrence of a CV hospitalization
  3. HF medication use and dose for i) an ACEi/ARB/ARNi, ii) a MRA, and iii) a beta-blocker
  Each participant in each comparison can have 0-8 points and all participants are compared using this score at the respective appropriate follow-up time point.
  RAASi=renin-angiotensin-aldosterone system inhibitor; ACEi=angiotensin converting enzyme inhibitor; ARB=angiotensin receptor blocker; ARNi=angiotensin receptor/neprilysin inhibitor; MRA=mineralocorticoid receptor antagonist.
Time Frame: Mean duration of exposure: 227.9 days for Patiromer and 234.5 days for Placebo
Measure: Number; unit: Events
Arm/Group | All Participants
Number analyzed (Participants) | 878
Events
  Number of wins in Patiromer Group | 62073
  Number of wins in Placebo Group | 49733
  Number of ties | 80915
  Total number of pairs | 192721
Statistical Analysis 1: Comparison: All Participants; Win ratio for composite. Win ratio approach: Patients in the new treatment and control groups are formed into matched pairs based on their risk profiles. For each matched pair, the new treatment patient is labelled winner/loser depending on CV/hyperkalemia event first. The win ratio is the total number of winners divided by the total numbers of losers. Unmatched win ratio is presented for this endpoint. Win ratio above 1 favors patiromer; Test type: Superiority; p = 0.048, Win Ratio; Win Ratio = 1.248, 95% CI 2-sided [1.003 to 1.564]

ADVERSE EVENTS:
Time Frame: Mean duration of exposure: 227.9 days for Patiromer and 234.5 days for Placebo
Arm/Group | Patiromer | Placebo
All-Cause Mortality (participants affected / at risk) | 24/439 | 18/439
Serious Adverse Events (participants affected / at risk) | 54/439 | 58/439
Other Adverse Events (participants affected / at risk) | 320/439 | 325/439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patiromer (N=439) | Placebo (N=439)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sudden death (General disorders) | 10 (10) | 10 (10)
Death (General disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ultrasound pancreas abnormal (Investigations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 9 (10) | 15 (18)
Angina unstable (Cardiac disorders) | 3 (3) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 4 (6)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 2 (2)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patiromer (N=439) | Placebo (N=439)
Hypotension (Vascular disorders) | 15 (17) | 13 (14)
Hypertension (Vascular disorders) | 8 (8) | 2 (2)
Asthenia (General disorders) | 5 (5) | 8 (9)
Oedema peripheral (General disorders) | 2 (2) | 5 (5)
Gynaecomastia (Reproductive system and breast disorders) | 6 (6) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 15 (19) | 10 (14)
Blood creatinine increased (Investigations) | 2 (2) | 5 (5)
Cardiac failure (Cardiac disorders) | 10 (11) | 10 (11)
Atrial fibrillation (Cardiac disorders) | 5 (6) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 5 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (9) | 7 (7)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (7)
Headache (Nervous system disorders) | 9 (9) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 19 (20) | 15 (15)
Constipation (Gastrointestinal disorders) | 11 (13) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 5 (7) | 8 (8)
Renal impairment (Renal and urinary disorders) | 5 (5) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 197 (335) | 238 (412)
Hypokalaemia (Metabolism and nutrition disorders) | 66 (75) | 47 (53)
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 (20) | 22 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (11) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Iron deficiency (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Pneumonia (Infections and infestations) | 7 (8) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 6 (8)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03888066/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT03888066/SAP_001.pdf